CLINICAL TRIAL: NCT03296163
Title: A Randomized, Multicenter, Multinational, Double-Blind Study to Assess the Efficacy and Safety of MB02 (Bevacizumab Biosimilar Drug) Versus Avastin® in Combination With Carboplatin and Paclitaxel for the Treatment of Subjects With Stage IIIB/IV Non-squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study Comparing MB02 and Avastin® in Subjects With Stage IIIB/IV Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Acronym: STELLA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB02-C-02-17
Record Dates: First submitted 2017-09-19; First posted 2017-09-28 (Actual); Results first posted 2021-03-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MB02 (Bevacizumab Biosimilar Drug) (Experimental): MB02 (Bevacizumab Biosimilar Drug) + Carboplatin/Paclitaxel
  Interventions: Drug: MB02 (Bevacizumab Biosimilar Drug); Drug: Carboplatin; Drug: Paclitaxel
- EU-approved Avastin® (Active Comparator): EU-approved Avastin® + Carboplatin/Paclitaxel
  Interventions: Drug: EU-approved Avastin®; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: MB02 (Bevacizumab Biosimilar Drug) — 15 mg/kg IV every 3 weeks on Day 1
  Other Names: Bevacizumab
  Arms: MB02 (Bevacizumab Biosimilar Drug)
Drug: EU-approved Avastin® — 15 mg/kg IV every 3 weeks on Day 1
  Other Names: Bevacizumab
  Arms: EU-approved Avastin®
Drug: Carboplatin — Carboplatin Area under the curve (AUC) 6 IV every 3 weeks on Day 1 for 6 cycles
Drug: Paclitaxel — Paclitaxel 200 mg/m2 IV every 3 weeks on Day 1 for 6 cycles
  Other Names: Taxol

SUMMARY:
This is a multicenter, multinational, double-blind, 1:1 randomized, parallel-group, equivalence Phase 3 study to compare the efficacy and safety of MB02 plus chemotherapy (carboplatin and paclitaxel) versus Avastin® plus chemotherapy (carboplatin and paclitaxel) in subjects with Stage IIIB/IV non-squamous NSCLC

DETAILED DESCRIPTION:
Efficacy parameters, safety profiles and immunogenicity will be compared between MB02 (Bevacizumab Biosimilar Drug) and European (EU)-approved Avastin®

ELIGIBILITY:
Inclusion Criteria:

1. Males and female subjects aged ≤ 18 years to ≤ 80 years.
2. Signed informed consent must be obtained before initiation of any study-specific procedures or treatment as confirmation of the subject's awareness and willingness to comply with the study requirements.
3. Subjects should have newly diagnosed or recurrent Stage IIIB/IV (defined by seventh edition of the Tumor, Node and Metastasis (TNM) classification for Lung Cancer, 2010) non-squamous NSCLC not amenable to curative intent surgery, and not have received any systemic therapy for advanced disease (exclusion criteria 3 and 4). For subjects with recurrent disease, at least 6 months must have elapsed before randomization from previous adjuvant treatment.
4. Previous radiation therapy if completed >4 weeks before randomization. Palliative radiotherapy to bone lesions is allowed if completed >2 weeks of randomization.
5. Subjects must have at least 1 unidimensional measurable lesion per RECIST version 1.1 (assessed locally).
6. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤1 at Screening.
7. Subjects must have adequate hepatic, renal and hematologic function defined as:

   * Hepatic function: bilirubin level <1.5 the upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels<2.5×ULN.
   * Renal function: serum creatinine level <1.5×ULN, calculated creatinine clearance (CrCl) >50 mL/min (Cockcroft-Gault formula), urine protein to creatinine ratio <1. Subjects with urine protein-to-creatinine ratio >1 may be enrolled if they have <1 g of protein in 24-hour urine collection.
   * Hematological function: Absolute neutrophil count >1.5×109 /L; platelets >100×109 /L, hemoglobin (Hb) >9 g/dL.
   * Adequate coagulation parameters such as: INR ≤ 2.0 and aPTT ≤ 1.5 x ULN within 7 days prior to randomization for patients not receiving anticoagulation therapy.
8. Eligible subjects must have a systolic blood pressure of ≤ 140 mm Hg and a diastolic blood pressure of ≤90 mm Hg at screening.
9. Women of childbearing potential, and their partners, must agree to adhere to pregnancy prevention methods throughout the duration of the study (including the Follow-up visits, where applicable). Women of childbearing potential are defined as those who are not surgically sterile (did not underwent bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) and not postmenopausal.

Subjects and their partners must agree to use a highly effective method of contraception, to avoid women becoming pregnant throughout the course of the study. Medically acceptable forms of birth control can include the following, with approval of the treating physician:

* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, sexual abstinence.

  10. Non fertile women can be included, that is, those who are physiologically incapable of becoming pregnant, because of:
* Hysterectomy.
* Bilateral oophorectomy (ovariectomy).
* Bilateral tubal ligation or,
* Postmenopausal women defined as:

Subjects not using hormone replacement therapy (HRT) and have experienced total cessation of menses for ≥ 1 year and be greater than 45 years of age, OR, in questionable cases, have a follicle stimulating hormone >40 mIU/mL and an estradiol value <40 pg/mL (<140 pmol/L).

Subjects must discontinue HRT before study enrolment because of the potential for inhibition of cytochrome enzymes that metabolize estrogens and progestins. For most forms of HRT, at least 2 to 4 weeks must elapse between the cessation of HRT and determination of menopausal status; the length of this interval depends on the type and dosage of HRT.

If a female subject is determined not to be postmenopausal, that subject must use adequate contraception, as defined immediately above (inclusion 8).

Exclusion Criteria:

1. Inability to comply with protocol procedures.
2. Participation in another clinical trial or treatment with another investigational agent within 4 weeks or 5 half-lives of investigational agent before randomization, whichever is longer.
3. Subjects previously treated with monoclonal antibodies or small molecule inhibitors against Vascular Endothelial Growth Factor (VEGF) or VEGF receptors, including Avastin®.
4. Subjects who have received previous chemotherapy, immunotherapy, targeted therapy, or biological therapy for their lung cancer. Note: Adjuvant and neo- adjuvant therapy are permitted (see: inclusion criterion 3).
5. Subjects who have known central nervous system disease, with the exception of subjects with treated brain metastases who have completed treatment (radiation, surgery or stereotactic surgery) and have not received steroids for at least 4 weeks before randomization. Subjects with central nervous system metastases treated by neurosurgical resection or brain biopsy performed within 8 weeks before randomization will be excluded. Subjects with known or history of brain metastases must undergo brain imaging during screening.
6. Current or recent (within 10 days of the first dose of study treatment) use of aspirin (at least 325 mg/day) or other nonsteroidal anti-inflammatory drugs with antiplatelet activity or treatment with dipyridamole (Persantine®), ticlopidine (Ticlid®), clopidogrel (Plavix®), or cilostazol (Pletal®).
7. Current or recent (within 5 days) use of therapeutic anticoagulation or use of thrombolytic agent. Prophylactic use of low molecular weight heparin is allowed.
8. Subjects with an INR >2, unless receiving active anticoagulation treatment, will be excluded.
9. Subjects who have a diagnosis of small cell carcinoma of the lung or squamous cell carcinoma of the lung. Mixed tumors should be categorized according to the predominant histology. If small cell elements are present, the subject will be excluded.
10. Subjects with known tumors that harbor activating epidermal growth factor receptor and anaplastic lymphoma receptor tyrosine kinase (assessed locally).
11. Subjects who have a history of hypersensitivity to the active substance (bevacizumab, carboplatin, and/or paclitaxel) or any of the excipients (such as trehalose dehydrate, sodium phosphate, or polysorbate 20).
12. Subjects with known active viral infection, including but not limited to: hepatitis B, hepatitis C, or HIV.
13. Subjects who are pregnant or breastfeeding. Women of child-bearing potential must have a negative pregnancy test at Screening.
14. Subjects with previous major surgery, open biopsy, open pleurodesis, or significant traumatic injury within 4 weeks before randomization or those anticipated to require major surgery during the study.
15. Subjects who have had a core biopsy taken or have had another minor surgical procedure, excluding placement of vascular access device, closed pleurodesis, thoracentesis, and mediastinoscopy, within 1 week of randomization.
16. Subjects with a history of abdominal fistula, GI perforation, intra-abdominal abscess within 6 months of randomization.
17. Subjects with a nonhealing wound, active ulcer, or untreated bone fracture.
18. Subjects with previous history of hypertensive crisis or hypertensive encephalopathy.
19. Subjects with New York Heart Association Grade II or greater congestive heart failure, or angina, myocardial infarction within 6 months before randomization; symptomatic arrhythmia or serious cardiac arrhythmia requiring medication; abnormal left ventricular ejection fraction < 50% assessed by ultrasound or multigated acquisition scan.
20. Subjects with a previous malignancy within 3 years of randomization (other than superficial basal cell and superficial squamous (skin) cell carcinoma, or carcinoma in situ of the uterine cervix, bladder, or prostate).
21. Subjects with history of a significant vascular event within 6 months before randomization (including, but not limited to myocardial infarction and stroke or transient ischemic attack).
22. Subjects with known bleeding diathesis or significant coagulopathy defined as a bleeding event grade ≥ 2 within 3 months before randomization.
23. Subjects with history of grade ≥2 hemoptysis within 6 months before randomization (≥0.5 teaspoons of bright red blood per event).
24. Subjects with a tumor(s) invading or compressing major blood vessels.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (118):
- Brazil (15):
  - MedRadius, Maceió, Alagoas
  - Instituto do Câncer do Ceará - ICC, Fortaleza, Ceará
  - Centro Brasileiro de Radioterapia Oncologia e Mastologia, Goiânia, Goiás
  - Hospital Erasto Gaertner - Paranaense de Combate ao Câncer, Curitiba, Paraná
  - Instituto Nacional de Cancer- INCA, Rio de Janeiro, Rio de Janeiro
  - Centro de Pesquisa e Educação da Serra Gaúcha (CEPESG), Caxias do Sul, Rio Grande do Sul
  - IPCEM Universidade de Caxias Do Sul, Caxias do Sul, Rio Grande do Sul
  - Hospital de Caridade de Ijuí, Ijuí, Rio Grande do Sul
  - Instituto do Câncer - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Pôrto Alegre, Rio Grande do Sul
  - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Hospital de Base de São José do Rio Preto, São José Do Rio Prêto, São Paulo
  - Centro de Pesquisa do Instituto Brasileiro de Controle do Câncer - IBCC, São Paulo, São Paulo
  - Instituto de Ensino e Pesquisa São Lucas, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo
- Bulgaria (3):
  - Central Hospital Plovdiv, Plovdiv
  - Acıbadem City Clinic Cancer Center UMHAT, Sofia
  - Specialized Hospital for Active Treatment of Oncology Diseases Sofia District EOOD, Sofia
- Chile (4):
  - Fundación Arturo López Pérez - Instituto Oncológico FALP, Santiago
  - Health & Care Spa, Santiago
  - Instituto Clinico Oncologico del Sur ICOS, Temuco
  - Oncocentro APYS, Viña del Mar
- Georgia (7):
  - Cancer Center of Adjara Autonomous Republic, Batumi
  - Acad. F . Todua medical center-research institute of clinical medicine, Tbilisi
  - Consilium Medulla, Tbilisi
  - Institute of Clinical Oncology, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - LTD Cancer Research Centre, Tbilisi
  - Tbilisi State Medical Universitys First university Clinic, Tbilisi
- Greece (5):
  - General Hospital of Athens "Ippokratio", Athens
  - Sotiria General Hospital for Chest Diseases, Athens
  - University General Hospital of Larissa, Larissa
  - Agioi Anargyroi General Oncological Hospital of Kifissia, Nea Kifissia
  - General Hospital of Thessaloniki "George Papanikolaou", Thessaloniki
- Hungary (5):
  - National Koranyi Institute of TB and Pulmonology, Budapest
  - Országos Korányi Pulmonológiai Intézet (OKPI), Budapest
  - Csongrád Megyei Önkormányzat Mellkasi Betegségek Szakkórháza, Deszk
  - Veszprém Megyei Tüdőgyógyinzézet, Farkasgyepű
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktatókórház, Miskolc
- India (14):
  - Zydus Hospital, Ahmedabad
  - Action Cancer Hospital, Delhi
  - Aadhar Health Institute, Hisar
  - NIMS - Nizam's Institute of Medical Sciences, Hyderabad
  - Ganadhipati Purushottam Shekhawati Hospital Research Centre, Jaipur
  - PVS Hospital Pvt Ltd, Kerola
  - Apollo Gleneagles Hospital, Kolkata
  - Netaji Subhas Chandra Bose Cancer Research Institute, Kolkata
  - Shatabdi Super Speciality Hospital, Nashik
  - Deenanath Mangeshkar Hospital & Research Center, Pune
  - Nirmal Hospital Pvt. Ltd., Surat
  - Kiran Super Multispeciality Hospital, Sūrat
  - Shree Himalaya Cancer Hospital Research Institute, Vadodara
  - Queen's NRI Hospital Gurudwara Lane, Visakhapatnam
- Notre Dame de Secours, Byblos, Lebanon
- Malaysia (7):
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Institut Perubatan dan Pergigian Termaju Universiti Sains Malaysia, Kepala Batas
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Pusat Perubatan Universiti Kebangsaan Malaysia, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
  - National Cancer Institute, Putrajaya
- Mexico (2):
  - Instituto Nacional de Cancerologia, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio González, Monterrey
- Sultan Qaboos University Hospital, Muscat, Oman
- Philippines (9):
  - Baguio General Hospital & Medical Center, Baguio City
  - Cebu Doctors University Hospital - CDUH, Cebu
  - Perpetual Succour Hospital - PSH, Cebu
  - St. Luke's Medical Center - Global City, City of Taguig
  - De La Salle University Medical Center - DLSUMC, Dasmariñas
  - Davao Doctors Hospital - DDH, Davao City
  - Makati Medical Center, Makati City
  - Philippine General Hospital - PGH, Manila
  - The Medical City, Pasig
- Russia (16):
  - SBHI Arkhangelsk Region - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk
  - Regional state budgetary Healthcare Institution "Belgorod oncology dispensary", Belgorod
  - State Budget Healthcare Institution Ivanovo Regional Oncology Dispensary, Ivanovo
  - Kaluga Regional Clinical Oncology center, Kaluga
  - Republic Clinical Oncology Dispensary, Kazan'
  - Kursk Republican Clinical Oncology Dispensary, Kursk
  - "VitaMed" LLC, Moscow
  - Moscow City Oncology Hospital No 62, Moscow
  - N. N. Blokhin Russian Cancer Research Center, Moscow
  - University Headache Clinic LLC, Moscow
  - GBUZ of SK Pyatigorsk Oncology Dispensary, Pyatigorsk
  - Ryazan Regional Clinical Oncology Dispensary, Ryazan
  - City Clinical Oncology Dispensary, Saint Petersburg
  - GUZ "Leningrad Regional Clinical Hospital", Saint Petersburg
  - State Budgetary healthcare Institution "Samara regional clinical oncology dispensary", Samara
  - Federal budget Healthcare Institution "Volga District Medical Centre" under Federal Medical and Biological Agency, Veliky Novgorod
- Serbia (5):
  - CHC Bezanijska Kosa, Belgrade
  - Institute of Oncology and Radiology of Serbia (IORS), Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
  - Clinical center Nis (Clinic for pulmonary diseases), Niš
- Hospital Universitario Puerta de Hierro Majadahonda, Madrid, Spain
- Thailand (5):
  - Bangkok International Hospital And Wattanosod Hospital, Bangkok
  - Chiang Mai University (CMU) - Maharaj Nakhon Chiang Mai Hospital Nakorn Chiang Mai Hospital, Chiang Mai
  - Chiang Rai Prachanukroh Hospital, Chiang Rai
  - Songklanagarind Hospital, Hat Yai
  - Buddhachinaraj Hospital, Phitsanulok
- Turkey (Türkiye) (2):
  - Istanbul Medeniyet University Medical Faculty, Istanbul
  - Suat Seren Chest Diseases Hospital, Izmir
- Ukraine (16):
  - Municipal Institution Cherkasy Regional Oncology Dispensary of Cherkasy Regional Council, Cherkasy
  - Public Higher Education Insititution of Ukraine "Bukovinian State Medical University", Chernivtsi
  - Clinical Oncology Dispensary, Dnipro
  - Multifield Clinical Hospital No.4, Dnipro
  - State Institution "Grigoriev Institute for Medical Radiology National Academy of Medical Science of Ukraine", Kharkiv
  - State Institution "V.T. Zaycev Institute of general and urgent surgery of National academy medical sciences of Ukraine", Kharkiv
  - Medical and Diagnostic Centre Private Enterprise of Private Manufacturing Company "ACINUS", Kropyvnytskyi
  - Municipal Institution "Kryviy Rih Oncology Dispensary" of Dnipropetrovsk Regional Council, Kryvyi Rih
  - National Cancer Institute, Kyiv
  - National Institute of Cancer, Kyiv
  - Healthcare facility "Volyn regional Oncological Dispensary", Lutsk
  - Lviv State Oncology Regional Treatment and Diagnostic Center, Lviv
  - Odessa Regional Clinical Oncology Dispensary, Odesa
  - Uzhgorod National University, Uzhhorod
  - Vinnytsia Regional Clinical Oncology Dispensary, Vinnytsia
  - Communal Institution "Zaporizhzhya Regional Clinical Oncological Dispensary" of Zaporizhzhya regional council, Zaporizhzhya

REFERENCES:
- [Derived] Trukhin D, Poddubskaya E, Andric Z, Makharadze T, Bellala RS, Charoentum C, Yanez Ruiz EP, Fulop A, Hyder Ali IA, Syrigos K, Katgi N, Lopez Chuken YA, Rumyana I, Reyes-Igama J, Costamilan RC, Del Campo Garcia A, Florez A, Paravisini A, Millan S; STELLA Investigators. Efficacy, Safety and Immunogenicity of MB02 (Bevacizumab Biosimilar) versus Reference Bevacizumab in Advanced Non-Small Cell Lung Cancer: A Randomized, Double-Blind, Phase III Study (STELLA). BioDrugs. 2021 Jul;35(4):429-444. doi: 10.1007/s40259-021-00483-w. Epub 2021 Apr 29. PMID 33914256

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 627 subjects were randomized and assigned to one of the study arms. Two subjects in the MB02 arm failed screening but were randomized in error. These subjects did not receive treatment. Another two subjects did not receive MB02 treatment due to death (one subject) and unacceptable toxicity (one subject).
  Two subjects in the European (EU)-approved bevacizumab did not receive study treatment due to investigator decision (one subject) and unacceptable toxicity (one subject).
Groups:
- MB02 (Bevacizumab Biosimilar Drug): MB02 (Bevacizumab Biosimilar Drug) + Carboplatin/Paclitaxel
  MB02 (Bevacizumab Biosimilar Drug): 15 mg/kg IV every 3 weeks on Day 1
  Carboplatin: Carboplatin AUC 6 IV every 3 weeks on Day 1 for 6 cycles
  Paclitaxel: Paclitaxel 200 mg/m2 IV every 3 weeks on Day 1 for 6 cycles
- EU-approved Avastin®: EU-approved Avastin® + Carboplatin/Paclitaxel
  EU-approved Avastin®: 15 mg/kg IV every 3 weeks on Day 1
  Carboplatin: Carboplatin AUC 6 IV every 3 weeks on Day 1 for 6 cycles
  Paclitaxel: Paclitaxel 200 mg/m2 IV every 3 weeks on Day 1 for 6 cycles
Period: Combination Therapy
Arm/Group | MB02 (Bevacizumab Biosimilar Drug) | EU-approved Avastin®
Started | 315 | 312
Completed | 207 | 220
Not Completed | 108 | 92
Period: Monotherapy
Arm/Group | MB02 (Bevacizumab Biosimilar Drug) | EU-approved Avastin®
Started | 207 | 220
Completed | 68 | 74
Not Completed | 139 | 146

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MB02 (Bevacizumab Biosimilar Drug) | EU-approved Avastin® | Total
Number analyzed (Participants) | 315 | 312 | 627
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.0 [54.0 to 67.0] | 61.0 [56.0 to 67.5] | 61.0 [55.0 to 67.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 122 | 244
  Male | 193 | 190 | 383
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 71 | 54 | 125
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 243 | 256 | 499
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Body surface area (BSA) [Median (Inter-Quartile Range); unit: m^2] | 1.780 [1.600 to 1.940] | 1.790 [1.595 to 1.940] | 1.780 [1.600 to 1.940]

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) at Week 18
Description: Objective response rate was assigned for a subject if the subject displayed either complete response (CR) or partial response (PR) per RECIST version 1.1 at Week 18, as assessed by independent radiological review committee (IRC).
  Overall Response (OR) = CR + PR.
Time Frame: 18 weeks from randomisation
Population: Primary efficacy analysis was done in the intention-to-treat (ITT) population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MB02 (Bevacizumab Biosimilar Drug) | EU-approved Avastin®
Number analyzed (Participants) | 315 | 312
Percentage of participants | 40.3 [34.9 to 46.0] | 44.6 [39.0 to 50.3]
Statistical Analysis 1: Comparison: MB02 (Bevacizumab Biosimilar Drug) vs EU-approved Avastin®; Test type: Equivalence — Equivalence analysis was based on the risk ratio (RR) (MB02/EU-approved Avastin) with an equivalence margin predefined [0.73, 1.36]. The ORR estimate was stratified using the Cochran-Mantel-Haenszel estimate of the RR and corresponding 2-sided 90% confidence interval (CI); Risk Ratio (RR) = 0.910, 90% CI 2-sided [0.780 to 1.060] — Direction of comparison is: For RR: MB02/EU-approved Avastin. 95% CI was also calculated: (0.758, 1.092)
Statistical Analysis 2: Comparison: MB02 (Bevacizumab Biosimilar Drug) vs EU-approved Avastin®; Test type: Equivalence — The ORR estimate was stratified using the Cochran-Mantel-Haenszel estimate of the risk difference (RD) (MB02-EU-approved Avastin) with an equivalence margin predefined [-12%, 12%] and corresponding 2-sided 95% CI; Risk Difference (RD) = -4.02, 90% CI 2-sided [-10.51 to 2.47] — Direction of comparison is: For RD: MB02 - EU-approved Avastin. 95% CI was also calculated: (-11.76, 3.71)

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was defined as the time from randomization to subsequent confirmed progression per RECIST version 1.1, or death (whichever occurred first), measured in weeks and months. For PFS assessment clinical progression (i.e., treatment discontinuation due to progression of disease) was also considered as an event.
Time Frame: At Week 52 from randomisation
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MB02 (Bevacizumab Biosimilar Drug) | EU-approved Avastin®
Number analyzed (Participants) | 315 | 312
weeks | 36.0 [33.0 to 36.43] | 37.3 [36.14 to 45.14]
Statistical Analysis 1: Comparison: MB02 (Bevacizumab Biosimilar Drug) vs EU-approved Avastin®; Test type: Other — Hazard ratio of MB02 versus EU-approved Avastin; a hazard ratio =1 indicated no difference in progressive disease(PD)/death between 2 reporting groups; >1 indicated an increase in PD/death in MB02; <1 indicated an increase in PD/death in EU-approved Avastin; Hazard Ratio (HR) = 1.187, 95% CI 2-sided [0.98 to 1.44]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization to subsequent death, measured in weeks and months.
Time Frame: At Week 52 from randomisation
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MB02 (Bevacizumab Biosimilar Drug) | EU-approved Avastin®
Number analyzed (Participants) | 315 | 312
weeks | NA [NA to NA] — NA: insufficient number of participants with events | NA [NA to NA] — NA: insufficient number of participants with events
Statistical Analysis 1: Comparison: MB02 (Bevacizumab Biosimilar Drug) vs EU-approved Avastin®; Test type: Other; Hazard Ratio (HR) = 1.108, 95% CI 2-sided [0.827 to 1.485]

4. Secondary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs)
Description: Comparison of Safety profile. Safety was monitored by incidence of adverse events (AEs). AEs were coded as per MedDRA (version 20.1) and severity was graded according to NCI-CTCAE (version 4.03);
Time Frame: Week 1 to week 52
Population: Safety analyses were performed in the Safety population, which consisted of all subjects who received at least 1 administration of investigational medicinal product.
Measure: Number; unit: participants
Arm/Group | MB02 (Bevacizumab Biosimilar Drug) | EU-approved Avastin®
Number analyzed (Participants) | 311 | 310
participants
  with ≥1 TEAE | 288 | 288
  with ≥1 Grade 3 or 4 TEAE | 131 | 125
  with ≥1 treatment-related TEAE | 264 | 270
  with ≥1 Grade 3 or 4 treatment-related TEAE | 98 | 91
  with at least one Serious TEAE | 58 | 54
  with ≥1 TEAE leading to discontinuation | 72 | 63
  with ≥1 treatment-related TEAE leading to discontinuation | 42 | 33

5. Secondary Outcome: Immunogenicity Assessments (Anti-drug Antibodies [ADA] and Neutralizing Antibodies [NAb])
Description: Incidence of anti-drug antibodies (ADA) and neutralizing ADAs (NAb). Analyses of ADA incidence rate, antibody titer, and neutralizing antibodies (NAb) (following the recommended 3-tier approach) were performed.
Time Frame: At Weeks 1, 4, 10, 19, 34 and 52 from randomization and, at the End of Treatment Visit if, an ADA sample has not been collected within the previous 3 weeks
Population: Immunogenicity was assessed in the Safety population.
Measure: Number; unit: participants
Arm/Group | MB02 (Bevacizumab Biosimilar Drug) | EU-approved Avastin®
Number analyzed (Participants) | 311 | 310
participants
  ADA positive | 53 | 50
  NAb positive | 10 | 13
  NO seroconversion | 239 | 247

ADVERSE EVENTS:
Time Frame: Throughout the study completion. An average of two years (from the beginning of the study at 06-February-2018 till last patient last visit in 27-February-2020).
Description: Coded according to Medical Dictionary for Regulatory Activities (version 20.1), and graded on the basis of the US National Cancer Institute's Common Terminology for Adverse Events (version 4.03). Table for "Other Adverse events" includes serious and non-serious events.
  Six (MB02: 4; EU-approved Avastin: 2) out of the 627 subjects randomized did not received treatment. Therefore, the "total number of participants at risk" comprised 621 subjects (MB02: 311 subjects; EU-approved Avastin:310).
Arm/Group | MB02 (Bevacizumab Biosimilar Drug) | EU-approved Avastin®
All-Cause Mortality (participants affected / at risk) | 23/311 | 24/310
Serious Adverse Events (participants affected / at risk) | 58/311 | 54/310
Other Adverse Events (participants affected / at risk) | 288/311 | 288/310
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MB02 (Bevacizumab Biosimilar Drug) (N=311) | EU-approved Avastin® (N=310)
Pneumonia (Infections and infestations) | 8 | 8
Empyema (Infections and infestations) | 3 | 0
Gastroenteritis (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 2 | 0
Brain abscess (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 7
Neutropenia (Blood and lymphatic system disorders) | 3 | 6
Anemia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 6
Pyrexia (General disorders) | 2 | 1
Asthenia (General disorders) | 0 | 2
Death (General disorders) | 2 | 0
Fatigue (General disorders) | 0 | 2
Sudden death (General disorders) | 2 | 0
Disease progression (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Hemorrhage intracranial (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Ischemic stroke (Nervous system disorders) | 1 | 1
Ataxia (Nervous system disorders) | 0 | 1
Cerebral ischemia (Nervous system disorders) | 1 | 0
Dysmetria (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Vision blurred (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MB02 (Bevacizumab Biosimilar Drug) (N=311) | EU-approved Avastin® (N=310)
Alopecia (Skin and subcutaneous tissue disorders) | 155 | 163
Anemia (Blood and lymphatic system disorders) | 101 | 94
Thrombocytopenia (Blood and lymphatic system disorders) | 41 | 42
Neutropenia (Blood and lymphatic system disorders) | 34 | 45
Leukopenia (Blood and lymphatic system disorders) | 24 | 18
Neuropathy peripheral (Nervous system disorders) | 38 | 41
Peripheral sensory neuropathy (Nervous system disorders) | 22 | 23
Paresthesia (Nervous system disorders) | 21 | 13
Fatigue (General disorders) | 39 | 36
Asthenia (General disorders) | 39 | 29
General physical health deterioration (General disorders) | 23 | 29
Weight decreased (Investigations) | 23 | 27
Platelet count decreased (Investigations) | 26 | 19
Alanine aminotransferase increased (Investigations) | 15 | 21
Aspartate aminotransferase increased (Investigations) | 14 | 22
Neutrophil count decreased (Investigations) | 18 | 18
Nausea (Gastrointestinal disorders) | 47 | 44
Diarrhea (Gastrointestinal disorders) | 29 | 27
Vomiting (Gastrointestinal disorders) | 22 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 20
Respiratory tract infection viral (Infections and infestations) | 16 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 22
Decreased appetite (Metabolism and nutrition disorders) | 14 | 20
Hypertension (Vascular disorders) | 24 | 26
Proteinuria (Renal and urinary disorders) | 18 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT03296163/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT03296163/SAP_001.pdf